CLINICAL TRIAL: NCT04988880
Title: Territorial Implementation and Evaluation of an Expert Patient Program to Improve the Empowerment and Quality of Life of People With Multiple Sclerosis
Brief Title: Territorial Implementation and Evaluation of a Multiple Sclerosis Expert Patient Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: PR(AG)334/2021
Record Dates: First submitted 2021-07-12; First posted 2021-08-04 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis; Quality of Life; Patient Empowerment; Patient Activation; Fatigue; Peer Group
Keywords: Peer Group; Multiple sclerosis; Patient Empowerment; Quality of life; Patient Activation; Fatigue
MeSH Terms: conditions — Multiple Sclerosis; Patient Participation; Fatigue

STUDY DESIGN:
Intervention Model Description: Pre-post intervention multicenter clinical study to evaluate the territorial implementation of a specific Multiple Sclerosis Expert Patient Program of Catalonia (PPEC-EM) based on peer learning regarding quality of life, knowledge and self-management related to the health process of participants in 6 areas in Catalonia. It will start after the approval of the respective CEICs. The deployment will consist of 12 groups of patients (2 per unit): 6 groups with people with recurrent MS and 6 with people with progressive MS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Relapsing multiple sclerosis group (Experimental): Multiple sclerosis relapsing groups: each unit will provide a group of participant with relapsing multiple sclerosis
  Interventions: Other: Multiple Sclerosis Expert Patient Program of Catalonia
- Progressive multiple sclerosis group (Experimental): Multiple sclerosis progressive groups: each unit will provide a group of participants with progressive multiple sclerosis
  Interventions: Other: Multiple Sclerosis Expert Patient Program of Catalonia

INTERVENTIONS:
Other: Multiple Sclerosis Expert Patient Program of Catalonia — It is intended to constitute 12 groups of patients (6 with relapsing and 6 for progressive MS; one of each type per unit). The study will be conducted virtually due to the current pandemic situation. Throughout 9 sessions (1 per week for 9 sessions), participants in the group will share knowledge and lived experiences on all aspects related to MS and their self-management. In each session there is a theoretical part to focus on the topic, conducted by the EP. Immediately afterwards, the EP will encourage interaction, facilitating the expression of doubts, questions or experiences about the contents. Its resolution will be sought among the group, resulting in empowerment and control over the health situation. The knowledge acquired will be based on the information provided by the EP and on the knowledge resulting from the life experiences regarding MS of all the people involved. In all sessions, a healthcare professional will act as an observer, providing help and support to the EP.
  Other Names: PPEC-EM

SUMMARY:
Introduction: Multiple sclerosis (MS) affects about 50,000 people in Spain, so it is essential to implement health interventions that meet their needs and demands. Expert patient programs facilitate health-related empowerment through peer learning. From a study of focus groups that identified the characteristics and contents of an expert patient program for MS and the ongoing pilot tests, the need for implementation in the different reference units of Catalonia is established.

Hypothesis: The territorial implementation in Catalonia of a Catalonia® Expert Patient Program for people with MS (PPEC-EM) based on peer learning will improve the quality of life, knowledge and self-management related to the health process of the participants.

Objective: To deploy and evaluate the territorial implementation of a PPEC-EM based on peer learning regarding the quality of life, knowledge and self-management related to the health process of the participants.

Methodology: Pre-post intervention multicenter clinical study. This study will begin after the approval of the respective Ethics Committees. The deployment will consist of 12 groups of patients (2 per unit): 6 groups with people with recurrent MS and 6 groups with people with progressive MS. A patient with MS previously trained by a team of health professionals will lead 9 educational group sessions (1 weekly session for 9 weeks) with 12 people with the same disease in order to improve the impact and self-management according to the health process. The main variable is the improvement of the quality of life and the secondary ones are the emotional impact, activation of the person, knowledge on the MS, fatigue, habits and lifestyles, use of the sanitary services and program-related experience of participants. All variables will be measured before and after the intervention and after 6 and 12 months. A pre-post comparability analysis will be developed in relation to the variables studied.

DETAILED DESCRIPTION:
Scope. The study will be carried out in 6 specialized reference units in Catalonia for the group of patients diagnosed with MS. All these units are multidisciplinary reference units in Girona, Barcelona, Tarragona and Lleida for the group of patients diagnosed or suspected of demyelinating disease and specifically MS.

Design. Pre-post intervention multicenter clinical study to evaluate the territorial implementation of a specific Multiple Sclerosis Expert Patient Program of Catalonia (PPEC-EM) based on peer learning regarding quality of life, knowledge and self-management related to the health process of participants in 6 areas in Catalonia. It will start after the approval of the respective Ethics Committees. The deployment will consist of 12 groups of patients (2 per unit): 6 groups with people with recurrent MS and 6 with people with progressive MS.

Population. All people with a diagnosis of MS treated in the 6 reference units of Catalonia for people with MS will be eligible to be recruited to participate in the deployment of the PPEC-EM.

Recruitment. The diagnosis and follow-up of patients is carried out in the respective units and involves therapeutic support by the multidisciplinary team in the clinical consultation, the day care clinic or through a spontaneous consultation. Once a clinical visit has been made by a healthcare professional, where lack of knowledge regarding MS or the need for support to perform an effective self-management are detected, patient will be referred to the centre's study coordinator to explain the study, its purpose and to provide complete information to the patient. In case of acceptance, the professional will assess whether IC / EC are met. If so, the study coordinator will ask participants for their informed consent.

Sample size. It is intended to constitute 12 groups of patients (6 for people with remitting and 6 for progressive MS; one of each type per unit). Based on the methodology used in the program, the recruitment target will be 12 subjects per group (144 individuals in total). This is expected to compensate for possible losses during the intervention to ensure a minimum presence of 8-10 subjects per group throughout the program (96-120 individuals).

Study variables Dependents: quality of life, emotional impact, fatigue, activation of the person, knowledge of MS, habits and lifestyles, use of health services (number of primary care visits; number of emergency department visits; number visits unscheduled in the MS unit), medication, nutrition, exercise and program-related experience of the EP and the participants.

Independent variables

* Sociodemographic: year of birth (YYYY); sex (woman / man); marital status (single / married or in a couple); family support (yes / no); level of education (no studies / basic / Professional Training-Baccalaureate / higher education); employment situation (student / active / retired - with a disability).
* Of the disease. Baseline. Date of diagnosis (DD / MM / YYYY); type of MS (recurrent / progressive); EDSS (X.X); family history of MS (yes / no); treatment (with MS treatment / no treatment); type of medication (self-administered / hospital-administered); name of the active ingredient; percentage of medication collected at a pharmacy or drug administered (XX.XX%).
* Of the disease. Follow-up. treatment (with MS treatment / no treatment); type of medication (self-administered / hospital-administered); name of the active ingredient; percentage of medication collected at a pharmacy or drug administered (XX.XX%); medication change during the program (yes / no); number of new relapses according to medical history (XX); EDSS (X.X).
* Program variables: Attendance at all program sessions (yes / no); number of sessions attended (0-9); attendance at session 1 (yes / no); attendance at session 2 (yes / no); attendance at session 3 (yes / no); attendance at session 4 (yes / no); attendance at session 5 (yes / no); attendance at session 6 (yes / no); attendance at session 7 (yes / no); attendance at session 8 (yes / no); attendance at session 9 (yes / no); attendance at the M6 follow-up session (yes / no); attendance at the M12 follow-up session (yes / no).

Description of the questionnaires and test

1. Quality of life. Multiple Sclerosis Quality of Live - 54 items (MSQoL-54) (Vickrey, Hays, Harooni, Myers, & Ellison, 1995) and its Spanish adaptation by Aymerich in 2006 (Aymerich et al., 2006). It is a self-administered questionnaire, filled in approximately 15 minutes. It consists of 54 items, 36 correspond to the generic SF-36 questionnaire and the remaining 18 are specific to MS. The items are distributed in 12 dimensions and 2 individual items that measure changes in health status (comparison between current health and previous year) and satisfaction with sexual function. In addition, two subtotals corresponding to two scales are obtained: mental and physical health. Therefore, the MSQoL54 questionnaire is a relevant tool for assessing the impact of the PPEC-EM on participants 'quality of life.
2. Emotional impact. The Hospital Anxiety and Depression Scale (HADS) (Zigmond & Snaith, 1983) and the Catalan version made by Soto in 2018 (Soto, Gras, & Planes, 2008) is a specific instrument for detecting the level of anxiety or depression of an individual in the last 7 days. It consists of a self-administered questionnaire of 14 items, 7 corresponding to the anxiety subscale and 7 to the depression subscale. Each of the items has a rating from 0 to 3 (0 being the minimum affectation and 3 the maximum). A score from 0 to 7 indicates no disorder, 8 to 10 is a questionable case, and ratings above 11 clearly indicate the presence of anxiety or depressive disorder respectively. For all this it is a useful tool to detect those individuals with a condition that would indicate the need for a referral to a health professional for assessment and care (exclusion criteria) and to evaluate the effectiveness of the program on MS-related emotional impact.
3. Cognitive impairment. The Brief International Cognitive Assessment for Multiple Sclerosis (BICAMS) battery was proposed in 2012 (Langdon et al., 2012) as a cognitive election screening tool in MS it is used widely internationally. It was translated into Spanish (Vanotti, Smerbeck, Benedict, & Caceres, 2016) and there are scales to determine whether a patient with MS has significant cognitive impairment. As described in the literature, if a patient has a score of -1.5 SD of the population mean in one of the 3 subtests administered, cognitive impairment is estimated. Patients who exceed this point will be excluded from the study.
4. Fatigue. The Fatigue Severity Scale (FSS) (Krupp, LaRocca, Muir-Nash, & Steinberg, 1989) and its Spanish translation by Tola in 1998 (Tola, Yugueros, Fernández-Buey, & Fernández-Herranz, 1998) is an instrument that assesses the impact of fatigue on a person's daily life. It consists of a self-administered questionnaire of 9 items, each with a rating from 1 to 7 (with 1 strongly disagreeing and 7 strongly disagreeing). Therefore, it will be possible to evaluate the impact of the program on the management of the fatigue of the participants.
5. Patient activation (engagement). The 13-item Patient Activation Measure (PAM-13) and its validation in Spanish by Moreno-Chico in 2017 (Moreno-Chico et al., 2017) is an instrument that assesses knowledge, skills and people's confidence in self-management of their health and medical care. It consists of a self-administered questionnaire of 13 items, each with a rating from 1 to 4 (with 1 strongly disagreeing and 4 strongly disagreeing). Therefore, it allows us to evaluate the impact of the program on the activation and involvement of the participants.
6. Knowledge of MS. The panel of experts of the PPEC developed a specific questionnaire about the knowledge of MS that includes information related to the disease and specific aspects identified by the target population through a study of focus groups (Robles-Sanchez et al., 2020) identified as essential to empower themselves regarding the health condition. This questionnaire will assess the impact of the program on the knowledge acquired.
7. Habits and lifestyles. The PPEC coordinating panel developed a specific questionnaire to assess habits and lifestyles, this questionnaire has already been used in other variants of the program demonstrating its usefulness in assessing changes due to participation in this program.
8. Socio-demographic and disease variables. The PPEC coordinating panel developed a specific questionnaire for each of these variables specifically for this study.
9. Patient Reported Experience. The panel of experts of the PPEC developed a specific questionnaire about the Patient Reported Experience that includes information related to the experience lived by individuals regarding the programme. This questionnaire will assess the experience of individuals regarding the intervention.

Data collection. All variables will be measured pre and post intervention and at 6 and 12 months, so a session will be held in these periods to collect the questionnaires and offer the possibility of clarifying concepts or doubts that may arise regarding the contents of previous sessions. Participants will receive the questionnaires to be filled in at their home by means of the corporate email of the program and these will be returned by the participants by e-mail. At 12 months after the study, the original questionnaires will be collected through a courier service by the PPEC-EM.

Intervention. The study will be conducted virtually due to the current pandemic situation (SARS-CoV-2). For this reason, Teams virtual platform will be used, provided by PPEC managers linked to the Generalitat de Catalunya and for use endorsed by the aforementioned institution. The aim of the intervention is to reinforce positive knowledge in a concise, clear way and with language that can be understood by the participants. (See intervention description for further information).

Analysis of results. Continuous variables will be described with mean and standard deviation (SD) or median and interquartile range (RIQ) in case of non-compliance with normality criteria and categorical variables with absolute frequency and percentages. The non-parametric U Mann-Whitney test for independent samples and the Wilcoxon test for dependent samples will be used to analyze the relationship between a category variable and a numerical variable. The Chi2 test or the Fisher's exact test will be used to analyze the relationship between two category variables. A significance level of 5% will be considered. The data will be analyzed using the SPSS statistical program with the latest version available.

Ethical aspects. The study protocol will be presented to the CEICs of the respective units. The foundations of the Declaration of Helsinki will be respected as well as the current legislation on confidentiality of personal data and the ethical norms on clinical studies, guaranteeing the strict fulfillment of the Law of protection of personal data, in Spain, Organic Law 3/2018, of 5 December, on the Protection of Personal Data and the guarantee of digital rights (BOE 6 December 2018, applicable from 7 December 2018). Participants will not be compensated for their inclusion or follow-up and will be informed of the voluntary nature of their participation, guaranteeing the confidentiality of data. All data collected will be incorporated into a computerized database, where participants will be identified with a code. No data will be shared. Each center will send the results to the HUVH coordinating center, the IP will guard the database. The database will be saved until the analysis is complete.

ELIGIBILITY:
Inclusion Criteria:

* Expert Patient: diagnosis of MS, possibility to attend the sessions and signing of the informed consent.
* Participants: Expert Patient inclusion criteria and need for support for self-management or detection of lack of knowledge regarding MS.

Exclusion Criteria:

* Expert Patient: not to speak or write Spanish or Catalan, healthcare or educational professional, having aphasia or an auditory disorder that prevents interaction with the group; -1.5 SD score of the population mean in one of the 3 subtests of The International Brief Cognitive Assessment for Multiple Sclerosis (BICAMS), score above 11/21 on The Hospital Anxiety and Depression Scale (HADS), and psychopathological comorbidity or diagnosed mental disorder that prevents proper interaction with the group.
* Participants: Expert Patient exclusion criteria without any restriction for healthcare or educational professionals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Number of groups constituted in each unit compared to the number of groups planned. | 18 months from recruitment
  Number of peer support groups provided by each centre. It is intended to develop two groups per unit (one group with progressive forms and one group with relapsing.remitting forms)

SECONDARY OUTCOMES:
Change in Quality of life measured by the Multiple Sclerosis Quality of Life 54 items (MSQOL54) from beginning of the intervention to end of intervention (9 weeks) and compared to 6 and 12 months after the end of the intervention. | 18 months from recruitment
  Multiple Sclerosis Quality of Live - 54 items (MSQoL-54) (Vickrey, Hays, Harooni, Myers, & Ellison, 1995) and its Spanish adaptation by Aymerich in 2006 (Aymerich et al., 2006). It is a self-administered questionnaire, filled in approximately 15 minutes. It consists of 54 items, 36 correspond to the generic SF-36 questionnaire and the remaining 18 are specific to MS. The items are distributed in 12 dimensions and 2 individual items that measure changes in health status (comparison between current health and previous year) and satisfaction with sexual function. In addition, two subtotals corresponding to two scales are obtained: mental and physical health.
Change in emotional impact measured by the Hospital Anxiety and Depression Scale (HADS) from beginning of the intervention to end of intervention (9 weeks) and compared to 6 and 12 months after the end of the intervention. | 18 months from recruitment
  The Hospital Anxiety and Depression Scale (HADS) (Zigmond & Snaith, 1983) and the Catalan version made by Soto in 2018 (Soto, Gras, & Planes, 2008) is a specific instrument for detecting the level of anxiety or depression of an individual in the last 7 days. It consists of a self-administered questionnaire of 14 items, 7 corresponding to the anxiety subscale and 7 to the depression subscale. Each of the items has a rating from 0 to 3 (0 being the minimum affectation and 3 the maximum). A score from 0 to 7 indicates no disorder, 8 to 10 is a questionable case, and ratings above 11 clearly indicate the presence of anxiety or depressive disorder respectively.
Change in fatigue management measured by the Fatigue Severity Scale (FSS) from beginning of the intervention to end of intervention (9 weeks) and compared to 6 and 12 months after the end of the intervention. | 18 months from recruitment
  The Fatigue Severity Scale (FSS) (Krupp, LaRocca, Muir-Nash, & Steinberg, 1989) and its Spanish translation by Tola in 1998 (Tola, Yugueros, Fernández-Buey, & Fernández-Herranz, 1998) is an instrument that assesses the impact of fatigue on a person's daily life. It consists of a self-administered questionnaire of 9 items, each with a rating from 1 to 7 (with 1 strongly disagreeing and 7 strongly disagreeing).
Change in patient activation and engagement measured by the 13-item Patient Activation Measure (PAM-13) from beginning of the intervention to end of intervention (9 weeks) and compared to 6 and 12 months after the end of the intervention. | 18 months from recruitment
  The 13-item Patient Activation Measure (PAM-13) and its validation in Spanish by Moreno-Chico in 2017 (Moreno-Chico et al., 2017) is an instrument that assesses knowledge, skills and people's confidence in self-management of their health and medical care. It consists of a self-administered questionnaire of 13 items, each with a rating from 1 to 4 (with 1 strongly disagreeing and 4 strongly disagreeing). The PAM-13 identifies four stages of activation of the individual.
Change in patient knowledge measured by the PPEC specific questionnaire about the MS knowledge from beginning of the intervention to end of intervention (9 weeks) and compared to 6 and 12 months after the end of the intervention. | 18 months from recruitment
  The panel of experts of the Expert Patient Program of Catalonia® (PPEC) developed a specific questionnaire about the knowledge of MS that includes information related to the disease and specific aspects identified by the target population through a study of focus groups (Robles-Sanchez et al., 2020) identified as essential to empower themselves regarding the health condition. This questionnaire will assess the impact of the program on the knowledge acquired.
Change in individuals habits and lifestyles measured by the PPEC specific questionnaire about the habits and lifestyles from beginning of the intervention to end of intervention (9 weeks) and compared to 6 and 12 months after the end of the intervention. | 18 months from recruitment
  The PPEC coordinating panel developed a specific questionnaire to assess habits and lifestyles, this questionnaire has already been used in other variants of the program demonstrating its usefulness in assessing changes due to participation in this program.
Change in the use of the care services from 1 year pre-intervention to end of intervention (9 weeks) compared to end of intervention (9 weeks) and 12 months after the end of the intervention. | 18 months from recruitment
  Use of health services according electronic clinical reports including number of primary care visits, number of emergency department visits, number visits unscheduled in the MS unit.
Change in Patient Reported Experience measured from the end of intervention (9 weeks) to 12 months after the end of the intervention. | 18 months from recruitment
  The panel of experts of the Expert Patient Program of Catalonia (PPEC) developed a specific questionnaire about the Patient Reported Experience that includes information related to the experience lived by individuals regarding the programme. This questionnaire will assess the experience of individuals regarding the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Angel Robles Sanchez, RN, Principal Investigator — Multiple Sclerosis Centre of Catalonia (Cemcat), Vall d'Hebron Barcelona Hospital Campus
Locations (6):
- Spain (6):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Centre d'Esclerosi Múltiple de Catalunya (Cemcat), Vall d'Hebron Barcelona Hospital Campus, Barcelona, Barcelona
  - Center for Neuroimmunology. Advanced Imaging in Neuroimmunological Diseases lab (ImaginEM). Hospital Clinic Barcelona, Barcelona, Barcelona
  - Unitat de Neuroimmunologia i Esclerosi Múltiple, Girona, Girona
  - Hospital Universitari Arnau de Vilanova Lleida; Institut de Recerca Biomèdica de Lleida (IRBLleida), Lleida, Lleida
  - Hospital Universitari de Tarragona Joan XXIII; Salut Sant Joan de Reus - Baix Camp; Fundació Esclerosi Múltiple - Mas Sabater, Tarragona, Tarragona

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.

REFERENCES:
- [Derived] Robles-Sanchez MA, Amil-Bujan P, Bosch-Farre C, Coll-Martinez C, Arevalo MJ, Anglada E, Menendez R, Montalban X, Sastre-Garriga J, Ramio-Torrenta L, Bertran-Noguer C. An expert patient program to improve the empowerment and quality of life of people with multiple sclerosis: protocol for a multicenter pre-post intervention study. Front Neurol. 2023 May 18;14:1172640. doi: 10.3389/fneur.2023.1172640. eCollection 2023. PMID 37273703